CLINICAL TRIAL: NCT02208999
Title: Two-years Follow-up of Post-spinal Implantable Neurostimulator PRECISION®
Brief Title: Follow-up of Post-spinal Implantable Neurostimulator PRECISION®
Acronym: PRECISION
Status: Completed | Type: Observational
Sponsor: Cemka-Eval (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011045; 913018 (Other: CNIL)
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Chronic Refractory Neuropathic Pain; Ischemic Peripheral Pain
Keywords: medullary neurostimulation; pain; Precision; rechargeable; implantable
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Neurostimulator Precision: Patients implanted or reimplanted with the neurostimulator Precision
  Interventions: Device: Neurostimulator Precision

INTERVENTIONS:
Device: Neurostimulator Precision — All patients included must have been implanted with the neurostimulator Precision

SUMMARY:
Assessing the long-term efficacy, complications, revision rates and final explantation of the device

DETAILED DESCRIPTION:
Longitudinal study with a follow-up of 2 years in patients implanted with the Precision neurostimulator.

This study will describe the characterisrics of the patients, of the implantation and will assess the long-term efficacy, complications, revision rates and final explantation of the device

ELIGIBILITY:
Inclusion Criteria:

* Adult patient receiving spinal implantation of a neurostimulator PRECISION ® ( primary implantation or reimplantation)

Exclusion Criteria:

* Refusal of patient
* Patient whose long-term monitoring will not be possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All implanted patients (primary implementation and reimplantation) with the neurostimulator PRECISION ®, during the inclusion period (1 year).
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Dr Mouton, MD, Study Director — Boston Scientific Corporation
Locations (1):
- Hospitals implanting the neurostimulator Precision, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; Only aggregated data will be communicated

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between December 3, 2015 and October 21, 2015 in 7 French clinical centers
Pre-assignment Details: No pre-assignment details
Groups:
- Patients Implanted or Reimplanted With Precision: All patients included must have been implanted with the neurostimulator Precision.107 patients were included. One of them was excluded because he was less than 18 years old. So 106 patients were analysed: 91 implanted patients (de novo implants) and 15 reimplanted patients (replacement implants)
Period: Overall Study
Arm/Group | Patients Implanted or Reimplanted With Precision
Started | 106
Completed | 105
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Implanted Patients: 91 patients de novo implanted with the neurostimulator Precision.
- Reimplanted Patients: 15 patients had a replacement with the neurostimulator Precision.
- Total: Total of all reporting groups
Arm/Group | Implanted Patients | Reimplanted Patients | Total
Number analyzed (Participants) | 91 | 15 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.0) | 51.7 (9.6) | 49.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 5 | 46
  Male | 50 | 10 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 91 | 15 | 106
Indication [Count of Participants; unit: Participants] — Type of pain for which the neurostimulator was implanted Population: 4 missing data
  Participants
    number analyzed (Participants) | 87 | 15 | 102
    Irreducible chronic neuropathic pain | 85 | 15 | 100
    Peripheral ischaemic pain | 2 | 0 | 2
Pain location [Count of Participants; unit: Participants] — Population: 1 missing data
  Participants
    number analyzed (Participants) | 90 | 15 | 105
    Unilateral pain | 56 | 5 | 61
    Bilateral pain | 34 | 10 | 44
Duration of pain before implant [Mean (Standard Deviation); unit: Months] — Mean age of pain (months) Population: 3 missing data
  Months
    number analyzed (Participants) | 88 | 15 | 103
    (all) | 68.0 (68.5) | 118.8 (101.6) | 75.4 (75.8)
History of pain surgery [Count of Participants; unit: Participants] — Population: 3 missing data
  Participants
    number analyzed (Participants) | 88 | 15 | 103
    (all) | 71 | 13 | 84
% of patients with a test phase before final implantation [Count of Participants; unit: Participants] — Population: 1 missing data
  Participants
    number analyzed (Participants) | 90 | 15 | 105
    (all) | 86 | 9 | 95
Percentage reduction in pain during the test phase [Mean (Standard Deviation); unit: percentage] — Population: 95 patients had a phase test and 4 data was missing.
  percentage
    number analyzed (Participants) | 83 | 8 | 91
    (all) | 69.2 (13.8) | 63.8 (11.9) | 68.8 (13.6)
Electrode insertion pathways [Count of Participants; unit: Participants] — Population: 1 missing data
  Participants
    number analyzed (Participants) | 90 | 15 | 105
    Percutaneous | 73 | 6 | 79
    Laminectomy | 16 | 8 | 24
    Percutaneous + laminectomy | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Implanted Patients (de Novo Implants) With an Improvement of at Least 50% of the Overall Average Pain Over the Last 8 Days, Evaluated by Numerical Scale at the First Follow-up Visit, at 1 Year, and 2 Years.
Description: Percentage of patients (de novo implants) having a reduction of usual pain over the past 8 days of at least 50% at 12 and 24 months. The pain was measured with a numerical scale from 0 to 10 (0 = no pain and 10 = most intense pain). This data has been provided by 71 patients at 1 year and by 70 patients at 2 years.
Time Frame: From baseline until the end of the study at 24 months.
Population: Implanted patients (de novo implants)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Implanted Patients (de Novo Implants): Primary outcome measure was estimated only in implanted patients (de novo implants)
Arm/Group | Implanted Patients (de Novo Implants)
Number analyzed (Participants) | 71
percentage of patients
  % patients with pain reduction >= 50% at &1 year | 34.5 [22.2 to 48.6]
  % patients with pain reduction >= 50% at 2 years: number analyzed (Participants) | 70
  % patients with pain reduction >= 50% at 2 years | 35.7 [24.6 to 48.1]

2. Secondary Outcome: Percentage of Implanted Patients (de Novo Implants) With an Improvement of at Least 30% of the Overall Average Pain, Evaluated by Numerical Scale
Description: Percentage of implanted patients (de novo implants) with an improvement of at least 30% at 12 and 24 months after inclusion for:
  * pain at the present time
  * usual pain over the past 8 days
  * the most severe pain in the last 8 days
Time Frame: From baseline until the end of the study at 24 months
Population: Percentage of de novo patients with an improvement of at least 30% for pain at 12 and 24 months after inclusion
Measure: Number (95% Confidence Interval); unit: % of patients
Groups:
- Implanted Patients (de Novo Implants) at 12 Months: Percentage of de novo patients with an improvement of at least 30% for pain at 12 months after inclusion
- Percentage of de Novo Patients at 24 Months: Percentage of de novo patients with an improvement of at least 30% for pain at 24 months after inclusion
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Percentage of de Novo Patients at 24 Months
Number analyzed (Participants) | 56 | 71
% of patients
  Pain at present time | 53.7 [39.6 to 67.4] | 53.6 [41.2 to 65.7]
  Usual pain over the past 8 days | 54.5 [40.6 to 68.0] | 51.4 [39.2 to 63.6]
  The most severe pain in the last 8 days | 46.3 [32.6 to 60.4] | 40.6 [28.9 to 53.1]

3. Secondary Outcome: Patients' Opinion on the Evolution of Pain
Description: - Pain relief compared to what the patient with a de novo implant, felt before the implantation at 12 months and at 24 months.
Time Frame: From baseline until the end of the study at 24 months
Population: Percentage of de novo patients for whom pain relief before the implantation was "improved" to "very improved" at 12 and 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Implanted Patients (de Novo Implants) at 12 Months: Percentage of de novo patients for whom pain relief before the implantation was "improved" to "very improved" at 12 months
- Percentage of de Novo Patients at 24 Months: Percentage of de novo patients for whom pain relief felt before the implantation was "improved" to "very improved" at 24 months
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Percentage of de Novo Patients at 24 Months
Number analyzed (Participants) | 54 | 70
Participants | 49 | 55

4. Secondary Outcome: Evolution of the Use of Other Pain Treatments
Description: Rate of primary implanted patients who took at least one analgesic treatment at each follow-up (at 1 year and at 2 years)
Time Frame: From baseline until the end of the study at 24 months
Population: Implanted patients (de novo implants) at 12 months and at 24 months with at least one analgesic treatment
Measure: Count of Participants; unit: Participants
Groups:
- Implanted Patients (de Novo Implants) at 12 Months: Rate of primary implanted patients who took at least one analgesic treatment at 1 year
- Percentage of de Novo Patients at 24 Months: Rate of primary implanted patients who took at least one analgesic treatment at 24 months.
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Percentage of de Novo Patients at 24 Months
Number analyzed (Participants) | 56 | 71
Participants | 42 | 54

5. Secondary Outcome: Evolution of Quality of Life (SF-12) - Physical Score
Description: Percentage of de novo patients with an increase of SF-12 (Short-Form health survey) physical score at 12 and 24 months. An increase of this score indicates an improvement in physical "quality of life.
Time Frame: From baseline until the end of the study at 24 months
Population: Percentage of de novo patients with an increase of SF-12 at 12 and 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Implanted Patients (de Novo Implants) at 12 Months: Percentage of de novo patients with an increase of SF-12 at 12 months
- Percentage of de Novo Patients at 24 Months: Percentage of de novo patients with an increase of SF-12 at 12 months at 24 months
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Percentage of de Novo Patients at 24 Months
Number analyzed (Participants) | 50 | 62
Participants | 30 | 38

6. Secondary Outcome: Patients' Willingness to Restart the Treatment
Description: Patients' willingness to restart the treatment at 12 months and at 24 months.
Time Frame: From baseline until the end of the study at 24 months
Population: Percentage of de novo patients willing to restart treatment at each follow-up (at 1 year and at 2 years)
Measure: Count of Participants; unit: Participants
Groups:
- Implanted Patients (de Novo Implants) at 12 Months: Percentage of de novo patients willing to restart treatment at 12 months
- Percentage of de Novo Patients at 24 Months: Percentage of de novo patients willing to restart treatment at 24 months
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Percentage of de Novo Patients at 24 Months
Number analyzed (Participants) | 49 | 66
Participants | 45 | 57

7. Secondary Outcome: Percentage of Patients With Anxiety and Depression Disorders
Description: Evolution of the rate of patients with anxiety and depression disorders at12 and 24 months.
Time Frame: From baseline until the end of the study at 24 months
Population: Percentage of de novo patients with anxiety and depression disorders at 12 and 24 months
Measure: Number (95% Confidence Interval); unit: percentage of included de novo patients
Groups:
- Implanted Patients (de Novo Implants) at 12 Months: Percentage of de novo patients with anxiety and depression at 12 months
- Percentage of de Novo Patients at 24 Months: Percentage of de novo patients with anxiety and depression at 24 months
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Percentage of de Novo Patients at 24 Months
Number analyzed (Participants) | 54 | 68
percentage of included de novo patients | 38.9 [27.6 to 52.8] | 45.6 [34.6 to 57.1]

8. Secondary Outcome: Evolution of Quality of Life (SF-12) - Mental Score
Description: Percentage of de novo patients with an increase of SF-12 (Short-Form health survey) mental score at 12 and 24 months. An increase of this score indicates an improvement in mental "quality of life.
Time Frame: From baseline until the end of the study at 24 months
Population: Percentage of de novo patients with an increase of SF-12 mental score at 12 and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Percentage of de Novo Patients at 24 Months
Number analyzed (Participants) | 50 | 62
Participants | 16 | 17

9. Primary Outcome: Average Pain Score Over the Last 8 Days, Evaluated by Numerical Scale at 1 Year, and at 2 Years.
Description: The pain was evaluated with a numerical scale from 0 to 10. 0 = no pain and 10 = most intense pain. This data has been provided by 71 patients at 1 year and by 70 patients at 2 years.
Time Frame: From baseline until the end of the study at 24 months.
Population: Implanted patients (de novo implants)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Implanted Patients (de Novo Implants)
Number analyzed (Participants) | 71
units on a scale
  Average pain score for the past 8 days at 1 year | 4.5 [2.2 to 6.8]
  Average pain score for the past 8 days at 2 years: number analyzed (Participants) | 70
  Average pain score for the past 8 days at 2 years | 4.9 [2.4 to 7.4]

10. Secondary Outcome: Evolution of the Use of Level 3 Analgesics
Description: Mean posology of level 3 analgesics at each follow-up (at 1 year and at 2 years). The posology was estimated in oral morphine equivalent dosage. At 1 year, 14 patients had a level 3 analgesic and at 2 years 18 patients had this type of analgesic. The posology was available for respectively 4 and 16 patients
Time Frame: From baseline until the end of the study at 24 months
Population: Implanted patients (de novo implants) at 12 months and at 24 months with at least one level 3 analgesic treatment
Measure: Mean (Standard Deviation); unit: MG
Groups:
- Implanted Patients (de Novo Implants) at 12 Months: Posology of level 3 analgesics at 12 months in de novo implanted patients
- Implanted Patients (de Novo Implants) at 24 Months: Posology of level 3 analgesics at 24 months in de novo implanted patients .
Arm/Group | Implanted Patients (de Novo Implants) at 12 Months | Implanted Patients (de Novo Implants) at 24 Months
Number analyzed (Participants) | 14 | 16
MG | 67.9 (55.4) | 55.6 (53.9)

ADVERSE EVENTS:
Time Frame: From baseline until the end of the study at 24 months
Description: Each investigator reported all adverse events from baseline until the end of the study at 24 months.
  The events were reviewed by an independent expert, who adjudicated whether each event was device related or not.
Groups:
- Overall Population: Implanted and Reimplanted Patients: Patients implanted (de novo implants) or reimplanted (replacement implants) with the neurostimulator Precision
- Patients With an Event Related to the Device: Patients implanted (de novo implants) or reimplanted (replacement implants) with the neurostimulator Precision and for whom the AE (or SAE) was related to this device
Arm/Group | Overall Population: Implanted and Reimplanted Patients | Patients With an Event Related to the Device
All-Cause Mortality (participants affected / at risk) | 2/106 | 0/106
Serious Adverse Events (participants affected / at risk) | 36/106 | 10/106
Other Adverse Events (participants affected / at risk) | 5/106 | 1/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Population: Implanted and Reimplanted Patients (N=106) | Patients With an Event Related to the Device (N=106)
Infections (Infections and infestations) | 8 (15) | 1 (1)
electrode displacement / electrode migration (Injury, poisoning and procedural complications) | 10 (11) | 1 (2)
Neurostimulator migration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Electrode fracture (Injury, poisoning and procedural complications) | 5 (6) | 5 (6)
Extension fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Undesirable stimulation (Injury, poisoning and procedural complications) | 5 (7) | 0 (0)
Loss of efficacy (Injury, poisoning and procedural complications) | 9 (11) | 1 (1)
Difficulty of charging (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Other complications (Injury, poisoning and procedural complications) | 11 (12) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Population: Implanted and Reimplanted Patients (N=106) | Patients With an Event Related to the Device (N=106)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Connector problem (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Undesirable stimulation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Loss of efficacy (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
High impedence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Study performed in real-life conditions , based on standard of care and some follow-ups were not considered as routine visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT02208999/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT02208999/SAP_001.pdf